CLINICAL TRIAL: NCT01580956
Title: Evaluation a New Ventilatory Modes: VARIABLE-PSV: a Randomized Controlled Cross-over Study: the " VARIABLE-PSV" Study
Brief Title: "VARIABLE-PSV" Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UF 8897
Record Dates: First submitted 2012-04-18; First posted 2012-04-19 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2012-04

CONDITIONS: Acute Respiratory Failure; Critical Illness; Ventilation Weaning
Keywords: Acute respiratory failure; Critical illness; Mechanical ventilation; Ventilation weaning; Intensive Care Unit; Variable (NOISY) PSV; PSV
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- VARIABLE-PSV ventilatory mode (Other)
  Interventions: Other: VARIABLE-PSV ventilatory mode
- STANDARD-PSV ventilatory mode (Other)
  Interventions: Other: STANDARD-PSV ventilatory mode

INTERVENTIONS:
Other: VARIABLE-PSV ventilatory mode — The two ventilatory modes will be studied during 24h in intubated patients in random order.
  Arms: VARIABLE-PSV ventilatory mode
Other: STANDARD-PSV ventilatory mode — The two ventilatory modes will be studied during 24h in intubated patients in random order.
  Arms: STANDARD-PSV ventilatory mode

SUMMARY:
Variable PSV is a new ventilatory mode which delivered a pressure support "variable" from 0 to 100% variation of the set PSV level.This study aimed to compare the ventilatory behavior, sleep quality and gas exchange between VARIABLE (or Noisy)-PSV and "standard" (or fixed)-PSV during the weaning phase of critically ill patients who required mechanical ventilation.

DETAILED DESCRIPTION:
Twenty patients will be enrolled. They will be ventilated withVARIABLE-PSV and STANDARD-PSV: for 24 h each in a randomized crossover order. The ventilatory parameters, ventilator/patient asynchrony, gas exchange effects, sleep quality and ventilatory comfort produced by the two ventilation modes will be compared. Before randomisation, a sequence of VARIABLE-PSV will be performed with different level of variation setting to better define the future behavior of the patient under this mode during the 24 h of Variable-PSV.

ELIGIBILITY:
Inclusion Criteria:

* ventilation planned for more than 48 h
* patient alert and calm corresponding to a Richmond Agitation-Sedation Scale (RASS) between -2 and 0
* Age > or equal 18
* Surrogate decision maker's consent

Exclusion Criteria:

* Clinical instability for any reason.
* Life support withdrawal code
* Patient under tutelage
* Pregnancy
* No French health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Oxygenation in each ventilatory mode | after 24h of mechanical ventilation in each mode
  We will performed arterial blood gases and oxygenation wil be evaluated by the PaO2/FiO2 ration.

SECONDARY OUTCOMES:
Ventilatory comfort | during 24h in each mode
  Comfort zone is defined as previously reported in some papers as considered adequate ventilation : 6 < tidal volume < 10 ml/kg, ETCO2 < 55 mmHg and < 65 mmHg for COPD patients and 12 < Respiratory rate < 35 cycles/min.
Feasibility | during the 24 hours
  Evaluation of time spent in each mode during the 24 hours of ventilation without any side effects and switch for another ventilatory mode.
Patient/ventilator asynchronism | during the 24 hours
  Evaluation of number of asynchrony evaluated by an Asynchrony Index (AI) in each mode during the 24 hours of mechanical ventilation
Ventilatory effects | during the 24 hours
  Evaluation of machine ventilatory behaviors in each mode during the 24 hours of mechanical ventilation.
Sleep quality | after the 24 hours
  Evaluation of quality of sleep in each mode after the 24h of mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology & Critical Care, St Eloi University Hospital, Montpellier, France